CLINICAL TRIAL: NCT05654012
Title: Migraine in Adolescents
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Hadas Nahman-Averbuch, Asst Prof of Anesthesiology, Washington University School of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 202208056; R01NS134986 (NIH); R01NS129742 (NIH)
Record Dates: First submitted 2022-11-28; First posted 2022-12-16 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — carboxypeptidase M; Efficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Family History of Migraine (Other): This group has a first degree relative diagnosed with migraine.
  Interventions: Device: MRI; Device: Thermal Stimuli; Device: Pressure stimuli; Behavioral: Pain ratings; Behavioral: Pressure pain thresholds (PPT); Behavioral: Conditioned pain modulation (CPM) efficiency; Diagnostic Test: Hormonal assessment; Behavioral: Migraine-related measures; Behavioral: Neural assessments; Diagnostic Test: Pubertal status
- No Family History of Migraine (Other): This group does not have a first or second degree relative diagnosed with migraine.
  Interventions: Device: MRI; Device: Thermal Stimuli; Device: Pressure stimuli; Behavioral: Pain ratings; Behavioral: Pressure pain thresholds (PPT); Behavioral: Conditioned pain modulation (CPM) efficiency; Diagnostic Test: Hormonal assessment; Behavioral: Migraine-related measures; Behavioral: Neural assessments; Diagnostic Test: Pubertal status

INTERVENTIONS:
Device: MRI — Grey Matter Volume (T1) Resting state BOLD
Device: Thermal Stimuli — The Thermal Sensory Analyzer (TSA-II or PATHWAY platform - Medoc, Ramat Yishai, Israel) will be used to safely deliver heat and cold stimuli. These devices can deliver relatively complex stimuli via computer control. All targeted stimulus temperatures will be less than 50°C, and participants will be free to remove their arm or leg at any time from the thermode. Noxious cold stimuli will also be delivered with a plastic water container or a water bath (FISHER, USA). Participants will be free to pull out of the water bath at any time.
Device: Pressure stimuli — Pressure stimuli will be applied by using a handheld algometer (Wagner Instruments) or the Pressure Algometer (Medoc, Ramat Yishai, Israel). These devices have a round probe that allows quantifying the amount of pressure that is being applied. The Pressure Algometer allows a real-time visual feedback to control and monitor applied pressure rates. Pressure will be applied to the lower leg, volar forearm, or trapezius.
Behavioral: Pain ratings — Pain intensity and pain unpleasantness ratings will be assessed by numerical rating scale (ranging from 0- no pain/unpleasantness to- 10 or 100 the most intense/unpleasantness pain imaginable) and by mechanical and computerized visual analog scales (VAS which ranges between ''no pain sensation'' and ''most intense pain imaginable'').
Behavioral: Pressure pain thresholds (PPT) — Pressure will be increased continually and participants will be instructed to press a button the first moment they feel pain from the pressure stimulus.
Behavioral: Conditioned pain modulation (CPM) efficiency — The CPM paradigm assesses endogenous inhibitory pain modulation efficiency related to spatial filtering of nociceptive information.
Diagnostic Test: Hormonal assessment — Blood samples will be collected for analyses of sex hormone levels
Behavioral: Migraine-related measures — Adolescents with migraine will complete questions regarding their headache frequency and migraine symptoms.
Behavioral: Neural assessments — MRI and fMRI scans
Diagnostic Test: Pubertal status — Pubertal status will be assessed using the self-reported Physical Developmental Scale-

SUMMARY:
Aim 1. To identify psychophysical and neural factors predicting migraine onset in adolescents

Aim 2a. To determine hormonal, psychophysical, and neural changes associated with migraine onset.

Aim 2b. To identify the temporal relationships between hormonal, psychophysical, and neural changes preceding vs. following migraine onset.

Aim 3. To identify psychophysical and neural factors predicting migraine prognosis in adolescents with migraine.

DETAILED DESCRIPTION:
This study aims to identify predictors of migraine onset in adolescents as well as to determine hormonal, psychophysical, and neural changes associated with migraine onset. The study procedures involve an MRI scan, sensory testing, blood draw, meeting with a specialist to determine migraine diagnosis, and completing surveys

After signing the consent/assent form, participants and their parent/legal guardian will complete surveys to ensure eligibility. At the beginning and/or after the baseline study visit and the beginning and/or after the follow-up study visits, participants will meet (in person or via electronic communication) with a headache/ pain specialist or a trained study staff member to determine if they meet the criteria for migraine diagnosis (based on the International Classification of Headache Disorders, 3rd Edition (ICHD-3) criteria). Participants will receive a copy of the Migraine Physician Meeting Summary Form (Migraine Summary Form). This may be sent to their email directly, email via DocuSign or in person at a study visit. For the healthy group, participants are required not to meet the criteria for migraine at the baseline study visit. For the migraine group, participants are required to meet the criteria for migraine diagnosis or present with migraine symptoms at the baseline study visit. Participants will be asked to complete a one-hour MRI scan and a psychophysical session which will include quantitative sensory testing (QST) assessments of pain sensitivity and inhibitory pain modulation capabilities (by testing the conditioned pain modulation response). During the psychophysical session, participants may also complete demographic, pubertal, and other surveys. At the end of the study visit, a blood draw may be conducted and a saliva sample might be collected for analyses of sex hormone levels. For two days following each study visit, participants may be asked to complete saliva samples, preferably at the same time as the study visit, to assess sex hormone levels. Additional blood and/or saliva samples may be collected at the study visits and stored for future genetic, hormonal or immune analyses.

Participants will complete short online monthly surveys for 2 years asking about the number of headaches in the last month, headache severity, causes for the headaches (e.g., virus), additional symptoms, and any new migraine diagnosis.

After 1 and 2 years, participants will return for follow-up study visits which may include the same procedures (MRI session, psychophysical session, completing surveys and a blood draw, and meeting with a headache/ pain specialist/trained study staff member).

Post menarche participants may have a pregnancy test before initiation of the study visit procedures. In case of pregnancy, participants will only meet with the headache/ pain specialist/trained study staff member and complete surveys. In addition, for post-menarche participants, if possible, the follow-up study visits may be scheduled at the follicular phase of the menstrual cycle (1-10 days after the beginning of menstruation).

If participants meet the diagnosis criteria for migraine at the follow-up study visits, they may be asked to complete additional surveys regarding their headaches characteristics (e.g., headache duration, intensity, and treatments, following the NINDS Common Data Elements,[2] and migraine-related disability which is widely used in pediatric patients.[43; 44] 28 days before and/or after the baseline and follow-up study visits, participants may be asked to complete a daily headache diary to assess headache frequency.

All study procedures are optional and participates can stop or not complete tests if they want.

ELIGIBILITY:
Inclusion criteria for healthy participants:

1. Age 10-13
2. Males or females (biological sex)
3. Not diagnosed with migraine or having migraine symptoms
4. With a first degree relative diagnosed with migraine (for the Fam-His group) or without a first or a second degree relative diagnosed with migraine (for the No-Fam-His group)

Inclusion criteria for participants with migraine:

1. Age 10-13
2. Males or females (biological sex)
3. Diagnosed with migraine or having migraine symptoms
4. Migraine duration > 6 months
5. Without preventative treatment or with stable preventative treatment for migraine (no change in intervention in the last 6 months)

Exclusion Criteria for the healthy group:

* Participants will not be enrolled if any of the following criteria exist and based on the investigator discretion:

  1. Diagnosis of any chronic pain syndrome
  2. Diagnosis of a neurological, developmental, pubertal, or psychiatric disorder
  3. Taking pain or psychiatric medications regularly
  4. Having an MRI contraindication such as metal in the body or claustrophobia
  5. Not able to understand and communicate in English

     Exclusion Criteria for the migraine group
* Participants will not be enrolled if any of the following criteria exist and based on the investigator discretion:

  1. Diagnosis of any chronic pain syndrome other than migraine
  2. Diagnosis of a neurological, developmental, pubertal, or psychiatric disorder
  3. Having an MRI contraindication such as metal in the body or claustrophobia
  4. Not able to understand and communicate in English

Ages: 10 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 250 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2028-03-15 (Estimated); Study Completion 2030-03-15 (Estimated)

PRIMARY OUTCOMES:
Number of participants with a new diagnosis of migraine | 2 years
  Multivariable regression analyses with baseline psychophysical, and neural factors will be used to identify predictors for migraine diagnosis and headache frequency.
  For Aim 1a, the primary outcome is migraine diagnosis (binary variable based on the physician's diagnosis), the independent variables are baseline PPT, CPM response, and FC of the right amygdala, and the controlling factors are race and age.
Number of participants with a new diagnosis of migraine | 2 Years
  Multivariable regression analyses with baseline psychophysical, and neural factors will be used to identify changes related to migraine diagnosis.
  For Aim 1b, the primary outcome measure is headache frequency (7-day average based on the headache diary completed before the 2-year follow-up visit), the independent variable is FC of the right amygdala, the controlling factors are the time of migraine diagnosis (at 1-year or 2-year study visit), race, and age. Since all participants will be at early pubertal maturation and pre-menarche at baseline, pubertal status will not be controlled for in this aim.

CONTACTS AND LOCATIONS:
Overall Officials: Hadas Nahman-Averbuch, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided